CLINICAL TRIAL: NCT07024355
Title: Predicting and Monitoring Spontaneous Bacterial Peritonitis in Cirrhotic Patients Using the Mansoura Scoring System
Acronym: MaSS/SBP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Principle Investigator, Assiut University
Other Study IDs: 04-2025-300593
Record Dates: First submitted 2025-04-23; First posted 2025-06-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-06

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective study was to examine predictors of SBP in order to develop a noninvasive method to identify or exclude an episode of SBP, for starting early treatment with antibiotics, so decrease morbidity and mortality in these patients.

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is a bacterial infection of ascitic fluid without any intra-abdominal, surgically treatable cause.

SBP is the most common bacterial infection in patients with cirrhosis, with a mortality rate exceeding 90% in untreated cases. However, inpatient mortality has been reduced to about 20% with early diagnosis and effective treatment.

Delayed diagnosis increases in-hospital mortality; with each hour of delay in performing paracentesis for SBP diagnosis, mortality increases by approximately 3.3%.

A study conducted in the United States reported that paracentesis was performed within the first 24 hours of admission in only 66% of cirrhotic patients with ascites.

Another study noted that routine paracentesis cannot be performed in all patients with liver cirrhosis. Therefore, delaying diagnosis increases mortality, and it is necessary to find a non-invasive and accurate method for predicting SBP.

Important risk factors for the development of SBP in cirrhotic patients include a history of SBP, variceal hemorrhage, and the use of proton pump inhibitors Several laboratory parameters have been evaluated as early predictors of SBP, including C-reactive protein (CRP), neutrophil-to-lymphocyte ratio (NLR), mean platelet volume (MPV), platelet count, and serum creatinine level. However, the data remain inconsistent.

Recently, the Mansoura Scoring System was developed at Mansoura University and retrospectively applied to cirrhotic patients with ascites for early SBP diagnosis without waiting for peritoneal fluid analysis.

The Mansoura score includes four components: age, MPV, and NLR (1 point each), and CRP (2 points), yielding a total score of 0 to 5. SBP is diagnosed when the score is equal to or greater than 4.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged >18 years
* Diagnosed liver cirrhosis
* Presence of ascites
* Provided written informed consent

Exclusion Criteria:

* Use of antibiotics within the previous two weeks
* Prophylactic treatment for spontaneous bacterial peritonitis (SBP) prior to admission
* Ascites not related to portal hypertension, including:
* Peritoneal tuberculosis
* Peritoneal carcinomatosis
* Congestive heart failure
* Renal disease
* Pancreatitis
* Hemorrhagic ascites
* Secondary peritonitis
* Presence of infections other than SBP, including:
* Pneumonia
* Urinary tract infection
* Skin and soft tissue infection
* Presence of malignancy Hematologic diseases
* Use of antiplatelet drugs or non-steroidal anti-inflammatory drugs (NSAIDs)
* Receipt of platelet or blood transfusion prior to admission
* Diseases associated with elevated mean platelet volume (MPV), including:
* Diabetes mellitus
* Cardiovascular disease
* Hyperthyroidism
* Immune thrombocytopenia
* Myeloproliferative disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This prospective study included all adult patients with cirrhosis and ascites admitted to AL-Rajhy Liver Hospital between April 2025 and April 2027
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the Mansoura Scoring System for Predicting Spontaneous Bacterial Peritonitis (SBP) | At hospital admission ( within 24 hours of admission)
  Primary Outcome Measure Title:Diagnostic Accuracy of the Mansoura Scoring System for Predicting Spontaneous Bacterial Peritonitis (SBP) Description: Evaluation of the diagnostic performance of the Mansoura scoring system in predicting spontaneous bacterial peritonitis (SBP), using ascitic fluid neutrophil count >250 cells/mm³ as the reference standard. Diagnostic accuracy will be assessed in terms of sensitivity, specificity, positive predictive value, negative predictive value, and area under the receiver operating characteristic (ROC) curve.
  Unit of Measure: Percentage / AUC

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Abdelmawgod, Lecturer, Trop Med, Principal Investigator — Assiut University